CLINICAL TRIAL: NCT06925347
Title: Comparıson Of The Effect Of Sılıcone And Acrylıc Medıcal Adhesıve Tapes On Skın İnjury In Fıxatıon Of The Nasogastrıc Tube
Brief Title: Comparıson Of Sılıcone And Acrylıc Medıcal Adhesıve Tapes On Skın İnjury Nasogastrıc Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ebru Ozel, Doctor Nurse, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: EGE-HMF-EO-01
Record Dates: First submitted 2025-03-16; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Medical-adhesive; Skin Injury
Keywords: nasogastric tube; medical-adhesive; silicone; acrylic; skin injury

STUDY DESIGN:
Intervention Model Description: It consists of 2 groups: control and experimental group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Medical adhesive tape with hypoallergenic acrylic adhesive used in standard practice was used in the control group (n=38).
  Interventions: Other: medical adhesive tape
- Experimental group (Experimental): Silicone medical adhesive tape was used in the experimental group (n=38).
  Interventions: Other: medical adhesive tape

INTERVENTIONS:
Other: medical adhesive tape — After the patients were assigned to the control and experimental groups, the tube of the patient in the control group was fixed with acrylic medical adhesive tape, and the tube of the patient in the experimental group was fixed with silicone medical adhesive tape.

SUMMARY:
This randomized controlled experimental study was conducted to compare the effects of silicone and acrylic medical adhesive tapes on medical-adhesive related skin injury in the fixation of nasogastric tubes in patients being monitored in intensive care.

DETAILED DESCRIPTION:
This randomized controlled experimental study was conducted to compare the effects of silicone and acrylic medical adhesive tapes on medical-adhesive related skin injury in the fixation of nasogastric tubes in patients being monitored in intensive care.

The population of the research consisted of patients with nasogastric tubes who were hospitalized in the Neurology Intensive Care Unit of Ege University Hospital (Health Practice and Research Center) between the dates of 01.06.2022 and 31.12.2023. The sample of the study consisted of 76 patients who were hospitalized in the Neurology Intensive Care Unit during this date range, had a nasogastric tube inserted, complied with the limitations of the study and agreed to participate in the study. Patients were stratified according to their age groups and assigned to experimental and control groups by block randomisation technique.

The nasogastric tube of the patients in the control group was fixed with acrylic medical adhesive tape which is used in routine practice, and the nasogastric tube of the patients in the experimental group was fixed with silicone medical adhesive tape. Starting from these condday following the nasogastric tube insertion, the medical adhesive tape that enables the fixation of the nasogastric tube was removed by wetting it with a sterile tampon impregnated with distilled water, and the patient's nasal skin was observed for 10 minutes each time, during 7 days for the presence of erythema, edema, denudation, dryness, infection, and vesicles. Then, the same medical adhesive tape was applied again and the tube was fixed. The data were analyzed in SPSS 25.0 program. Mann-Whitney U test, Pearson Chi-square test and Fisher's Exact probability test were used to analyze the data. The nasogastric tube of the patients in the control group was fixed with acrylic medical adhesive tape which is used in routine practice, and the nasogastric tube of the patients in the experimental group was fixed with silicone medical adhesive tape.

ELIGIBILITY:
Inclusion Criteria:

* Feeding with a nasogastric tube
* Being between the ages of 18-85
* Voluntarily participating in the study
* Having the first nasogastric tube inserted after admission to the Intensive Care Unit and having the tube detected by the researcher.

Exclusion Criteria:

* Having any dermatological disease
* Having a history of allergy
* Having a lesion on the skin of the nose
* Failure to detect the tube by the researcher when the first nasogastric tube was inserted after admission to the Intensive Care Unit.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Skin Evaluation Form | seven days
  Skin Assessment Form is a form developed by a dermatologist and researcher to evaluate whether there is skin injury on the nose skin of patients. The nose skin of patients was evaluated daily in terms of erythema, edema, denudation, dryness, infection, and vesicle presence and recorded on this form.

SECONDARY OUTCOMES:
Pain Assessment Form | seven days
  The Pain Assessment Form is a form used to determine the presence and severity of pain during the removal of medical adhesive tape from the patient's nose skin. The 3 different pain scales (numeric, facial and behavioral) routinely used in the intensive care unit where the study was conducted and the patient's pain score are included in this form

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Özel, Ph.D, Study Director — Ege University
Locations (1):
- Ege University Hospital (Health Practice and Research Center), Izmir, Bornova, Turkey (Türkiye)